CLINICAL TRIAL: NCT04543396
Title: Utilization of Tonal Exercise System to Improve Short- and Long-term Low Back Pain (LBP) Outcomes
Brief Title: Tonal Exercise System to Improve Short and Long Term Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aaron Krych, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-007281
Record Dates: First submitted 2020-08-27; First posted 2020-09-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain
Keywords: Tonal; low back pain; nonspecific; physical therapy; chiropractic; resistance training
MeSH Terms: conditions — Low Back Pain | interventions — Resistance Training; Timbre Perception

STUDY DESIGN:
Intervention Model Description: Four study groups will be assessed in parallel. Subjects will encompass patients who have sought physical therapy or chiropractic care for nonspecific lower back pain. Clinical care selection will be made by subject and clinical care team prior to study enrollment and will be made in the best interest of the subject. Intervention groups will consist of standard of care and an 8-week physical training supplement performed that will consist of concentric and eccentric resistance exercises as well as dynamic warm-up and cool-down periods. These interventions will be performed in addition to the standard regimen of clinical care.
Who Masked: Investigator
Masking Description: Investigator will be blinded to subject intervention group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical Thearpy + Resistance Training (Experimental): Subjects will receive standard of care treatments from their physical therapist. In addition, an investigative team member will customize a program of core-strengthening resistance exercises that will be prescribed to all intervention group subjects. Subjects will be expected to complete the protocol twice (2x) per week for an 8 week period. The protocol was approved by the Mayo Clinic IRB. Evaluations will be completed at baseline, week 4, and week 8 for all subject groups. Evaluations will consist of a strength assessment, standard clinical questionnaires about back health, a Sorenson's Back Endurance Test, and ultrasound images of back musculature. Longitudinal follow-ups will be completed quarterly for one year after the initial evaluation. These follow-ups will be performed remotely via phone and/or email and incorporate clinical questionnaires.
  Interventions: Other: Resistance exercise
- Physical Thearpy (No Intervention): Subjects will receive standard of care treatments from their physical therapist. Evaluations will be completed at baseline, week 4, and week 8 for all subject groups. Evaluations will consist of a strength assessment, standard clinical questionnaires about back health, a Sorenson's Back Endurance Test, and ultrasound images of back musculature. Longitudinal follow-ups will be completed quarterly for one year after the initial evaluation. These follow-ups will be performed remotely via phone and/or email and incorporate clinical questionnaires.
- Chiropractic Care + Resistance Training (Experimental): Subjects will receive standard of care treatments from their chiropractor. In addition, an investigative team member will customize a program of core-strengthening resistance exercises that will be prescribed to all intervention group subjects. Subjects will be expected to complete the protocol twice (2x) per week for an 8 week period. The protocol was approved by the Mayo Clinic IRB. Evaluations will be completed at baseline, week 4, and week 8 for all subject groups. Evaluations will consist of a strength assessment, standard clinical questionnaires about back health, a Sorenson's Back Endurance Test, and ultrasound images of back musculature. Longitudinal follow-ups will be completed quarterly for one year after the initial evaluation. These follow-ups will be performed remotely via phone and/or email and incorporate clinical questionnaires.
  Interventions: Other: Resistance exercise
- Chiropractic Care (No Intervention): Subjects will receive standard of care treatments from their chiropractor. Evaluations will be completed at baseline, week 4, and week 8 for all subject groups. Evaluations will consist of a strength assessment, standard clinical questionnaires about back health, a Sorenson's Back Endurance Test, and ultrasound images of back musculature. Longitudinal follow-ups will be completed quarterly for one year after the initial evaluation. These follow-ups will be performed remotely via phone and/or email and incorporate clinical questionnaires.

INTERVENTIONS:
Other: Resistance exercise — A training program designed to enhance core strength, stability, and function will be performed on the Tonal device. Training sessions will occur twice weekly for eight weeks. Performance of this program will be supervised by a designated and clinically trained research team member who will not conduct the statistical analysis and subsequently not be blinded to Group assignment. The program will last approximately 20 minutes in length and incorporate the a series of progressive exercises.
  Other Names: Tonal
  Arms: Chiropractic Care + Resistance Training; Physical Thearpy + Resistance Training

SUMMARY:
This study will assess the effect of incorporating a tonal exercise device into clinical and chiropractic care for lower back pain.

DETAILED DESCRIPTION:
All accrued subjects will be assigned study ID numbers to de-identify subject data and keep research team members blinded to group assignments. The CRC will maintain a master keyfile of subject Group randomization that will be revealed to the research team after between-group statistical analyses have been performed.

For all subjects: The active study period for this investigation will be 8 weeks in duration. Passive monitoring will then continue for 12 months after the initial 8 week period. All subjects will continue to receive standard of care treatments from their preferred clinical practitioner (physical therapist, chiropractor, none). All subjects will complete three progress assessments over the duration of the 8-week intervention period. These progress assessments will occur at baseline, week 4, and week 8 and will include the following elements:

1. Clinical Questionnaires - Clinical questionnaires will be digitally completed by each participant. There will be four (4) clinical questionnaires (Visual Analog Pain Scale, Tampa Scale for Kinesiophobia, PROMIS Physical Function, and PROMIS Pain Interference).

   PROMIS Physical Function Questionnaire: Developed by the NIH, this question bank is used to assess patient function. Patients rate each question on a nominal scale from 1-5 related to their ability to complete activities of daily living and exercise. We will use the version 2.0 question bank.

   PROMIS Pain Interference: Developed by the NIH, this question band is used to assess the degree to which pain interferes with quality of life and how much pain restricts the patient from activities of daily living and exercise. We will use the version 1.1 question bank.

   Tampa Scale for Kinesiophobia: Developed in 1990, this is a clinical questionnaire used to evaluate fear of movement relative to lower back pain. This is a 17 item form with each item being subjectively indicated by the subject on a 4 point scale. The overall form is then evaluated by a standardized scoring format.

   Visual Analog Scale: A one question clinical questionnaire that asks subjects to subjectively rate their pain on a scale from 1-10. A green-to-red color gradient may also be used and converted to a 10 point scale as this has shown to produce greater reliability.

   Patient Satisfaction: Subjects will be asked 2 questions related to satisfaction with their outcomes. Both questions will be scored on 5 point scales. Question 1 will be in reference to overall satisfaction "How would you rate your current satisfaction as related to your lower back pain?" Answer options will include 1) "very satisfied", 2) "somewhat satisfied", 3) "satisfied", 4) "somewhat dissatisfied", 5) "very dissatisfied". Question 2 comes from the North American Spine Society lumbar spine outcome assessment and will read "Rate your satisfaction of the treatment received for your lower back pain." Answer selections will include: 1) "The treatment met my expectations", 2) "I did not improve as much as I had hoped, but I would undergo the same treatment for the same outcome", 3) "I did not improve as much as I had hoped, and I would not undergo the same treatment for the same outcome", and 4) "I am the same or worse than before treatment".
2. Tonal Subject Satisfaction - Subjective questions pertaining to progress perceived by the subject will be integrated into the Tonal software platform and answers will be recorded digitally. The Tonal satisfaction question will be presented in the following format:

   Question for trial participants: "How was your workout?" Responses: 1, 2, 3, 4 or 5 stars

   If 1 star, the secondary question is: "Let's fix it. What can we improve?" If 2 - 4 stars, the secondary question is: "Thanks for your feedback. What can we improve?" If 5 stars, the secondary question is: "Thanks for your feedback. What did you love?"

   Selections:
   * Ease of use
   * Movements
   * Weight suggestions
   * Pacing
   * Results
   * Other (allows text to be entered freely)
3. Core Training Program - for intervention groups, a training program designed to enhance core strength, stability, and function will be performed on the Tonal device. Performance of this program will be supervised by a designated and clinically trained research team member who will not conduct the statistical analysis and subsequently not be blinded to Group assignment. Group 5 will also complete the prescribed training program in the comfort of their own home/Tonal gym. The program will last approximately 20 minutes in length and incorporate progressive exercises.

   Each training session will be preceded by a dynamic warm-up and finished with a dynamic cooldown to fit within the approximate time frame of 30 minutes. If at any point a prescribed exercise appears to cause difficulty or discomfort to a subject, the supervising trainer will have authority to use his/her discretion to modify the exercise to make it easier for the subject, or skip the exercise altogether. Throughout the training program, the Tonal device will record continuous data on range of motion, power generated, weight resistance, total weight displacement, time under tension, and strength score. This data is automatically saved on the Tonal servers and will be transferred to the research team on a weekly basis.

   At each evaluation session, subjects will perform the artificial intelligence learning program used by the Tonal to establish baseline resistance levels for new users. Subjects will be asked to perform five separate activities (neutral grip deadlift, bench press, overhead press, and lateral pull down), each for multiple repetitions. During the each repetition, the artificial intelligence program on the Tonal will adjust user resistance based on performance of the previous repetition until an optimal resistance weight is identified for the subject. Once the Tonal has established resistance levels, the subject will repeat each activity for 10 repetitions with weight activated. A weight-activated bicep curl will also be performed for 10 repetitions. The standard tonal data sheet will be collected. This sheet includes the following variables: activity, time, repetitions, range of motion, power, duration, target repetitions, target time, target duration, base weight, suggested weight, additional eccentric/concentric weight, assisted weight, total duration, total activities, total sets, total volume, and percent completion. Identifiable information, which is typically included in Tonal reports will be replaced with assigned Subject IDs prior to any data transfer so that all data remains de-identified. In addition to this standard Tonal report, continuous data will be collected for range of motion (calculated from cable distance traveled) and speed of motion relative to time.

   For each training session subjects will follow the specified exercise protocol, which will be supervised by the athletic trainer. The standard Tonal report will be generated as indicated for the evaluation sessions. This report will again be de-identified.
4. Sorenson's Back Endurance Test - a research team member will perform a Sorenson's Back Endurance Test on each subject. To perform this test, subject will lie prone on a clinical exam table with the superior edge of the iliac crest at the edge of the table and arms crossed over the chest. The lower limbs will be stabilized to the table with straps. The subject will be asked to maintain their upper body in a horizontal position for as long as possible while a research team member times them. If the subject maintains this posture for 240 seconds, the test will end. The total time for which a horizontal upper body posture is maintained will be recorded.
5. Shearwave Elastography (SWE) - SWE ultrasound images will be captured on the erector spinae muscles with a Aixplorer MACH 30 (Hologic Supersonic Imagine, France). This non-invasive, non-radiation imagery allows for assessment of stiffness properties in muscle tissue. A research team member will take SWE images with the subject laying prone on a horizontal surface in a relaxed position and with the ultrasound transducer aligned with the muscle fibers. A minimum of 3 images will be captured and averaged to determine the mean resting tissue stiffness. These ultrasound images are research procedures that will be completed by research staff using research equipment. The research team members have been trained in the collection of shearwave images directly by the ultrasound vendor company. The indicated activities will be completed supplemental to your standard clinical care as part of this study and will not be considered part of your medical treatment nor will they be included as part of your medical record.
6. Isokinetic Lumbar Strength - a research team member will assess flexion/extension torque of the lumbar spine will be assessed via a Humac Norm Dynamometer (CSMI Solutions, Stoughton, MA, USA). Isokinetic torque will be recorded across a subject-specified range of motion at a rotation speed of 60°/sec. A subject will be permitted four (4) warm-up trials to familiarize themselves with the isokinetic device and lumbar exercise. The subject will then be asked to perform five (5) recorded trials at their maximal effort.
7. Isometric Proprioceptive Measurement - a research team member will assess the ability of each subject to use their proprioception to match a target strength magnitude for isometric back flexion/extension contractions. This test will be performed using the lumbar accessory for the Humac Norm Dynamometer. A target force of will be selected. This test will be performed after the Isokinetic Lumbar Strength test and subjects will only qualify if their maximal isokinetic strength exceeds the specified target force. Subjects will be secured at a predetermined flexion angle within each subject's range of motion for lumbar flexion. Subjects will be asked to increase the strength of their back contraction in a trapezoidal form (3 seconds ramp-up, 10 seconds hold steady, 3 seconds ramp-down). The first trial will be performed with visual stimulus to define the target force. The second trial will be performed without visual stimulus and will rely on the subject's proprioception to identify the target force and maintain steadiness. These tests will be repeated three times.

For Standard of Care Subjects: Subjects will continue their preferred clinical care, but complete no additional Tonal training outside of the three progress evaluation sessions specified above.

For Intervention Subjects: Subjects will continue their preferred clinical care and additionally be asked to perform the above specified Core Training Program two (2) times per week for a period of eight (8) weeks. This program will be performed on a Tonal device installed at Mayo Clinic. For every training session, the Tonal Subject Satisfaction and Visual Analog Scale questions indicated above will be answered relative to the workout. Intervention subjects will complete a total of 16 training sessions on the Tonal device, with full progress evaluations occurring on sessions 1, 8, and 16.

Longitudinal Tracking: After the completion of the 8 week intervention period, all subjects from all Groups will be tracked by the CRC or research team members for up to one (1) year. The CRC or research team members will follow-up once per quarter with all subjects from all Groups. These follow-ups will be completed remotely via phone and/or email and will consist of quarterly interactions during which subjects will be asked to complete the same Clinical Questionnaires described above in the progress evaluations. Subjects will also indicate whether they have sought additional treatment for LBP. For Groups 1-4, those subjects that have had positive LBP recurrence will have their medical records evaluated for severity and outcome of LBP.

ELIGIBILITY:
Subjects seeking treatment for nonspecific LBP will be recruited by their treating therapist, physiatrist, athletic trainer, or chiropractor then enrolled by a clinical research coordinator (CRC). The CRC will assign study IDs and randomize clinical patients into groups based on the each subject's selected treatment of choice. Care will be taken to match subject distribution between groups based on demographics (sex and age), activity level, and subjective pain scores. Lead investigators will remain blinded to group assignments. Subjects will have to complete 2 screening evaluations prior to participation in this study. The first screen will be that the treating physical therapist, physiatrist, athletic trainer, or chiropractor will approve the patient for participation. The second screen will consist of completing two basic activities on the Tonal at minimal weight without being restricted by pain. The two activities will be 10 repetitions on each arm of standing unilateral bicep curl and seated unilateral lateral pulldown. For both activities Tonal resistance will be set at 5 pounds, which is the minimum resistance for the device. This screen will affirm that the subject is capable of completing at least the minimum level of workout provided by the Tonal.

Inclusion Criteria:

* Males and Females between ages 18 and 65
* Seeking physical therapy (PT) or chiropractic care
* Non-specific LBP
* Treatment at Mayo Clinic Rchester

Exclusion Criteria:

* Not able to attend Mayo Clinic Rochester for treatment
* Women who are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Patient Pain | 1 year
  Subjective assessment of patient pain scores as assessed by a 0-10 Visual Analog Scale, where 0 is no pain and 10 is the worst pain imaginable.
PROMIS Subjective Health Assessment score | 2 years
  Subjective assessment of patient health performed with the Patient-Reported Outcomes Measurement Information System (PROMIS) computer adaptive test. Scores range from 14.1-61.7 with higher scores representative of better functioning.
Kinesiophobia | 2 years
  Subjective assessment of patient fear of movement as assessed by the Tampa Scale of Kinesiophobia questionnaire. Scale is scored from 17-68 where higher scores indicate increased fear of movement.
Isometric Lumbar Strength | 1 year
  Maximum lumbar flexion/extension strength as determined with a Humac dynamometer isometric lumbar attachment.

SECONDARY OUTCOMES:
Frequency of Back Pain Recurrence | 2 years
  Number of recurrent visits and time between visits for low back pain that occur after completion of intervention period.
Functional Strength | 1 year
  Objective strength as assessed by Tonal artificial intelligence algorithm.
Lumbar Endurance | 1 year
  Time to lumbar muscle fatigue as determined by the Sorenson's Back Endurance Test

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Krych, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No